CLINICAL TRIAL: NCT01759004
Title: Muscle Strength and Physical Fitness in Patients With Lipedema and Obesity: a Prospective Cross-sectional Pilot Study
Brief Title: Physical Condition in Lipedema and Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nij Smellinghe Hosptial (Other)
Responsible Party: Principal Investigator, R.J. Damstra, Dermatologist MD PhD, Nij Smellinghe Hosptial
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NS4NL; Nij Smellinghe hospital (Other: Nij Smellinghe hospital)
Record Dates: First submitted 2012-12-04; First posted 2013-01-01 (Estimated); Last update posted 2013-12-06 (Estimated); Status verified 2013-12

CONDITIONS: Lipoedema; Obesity
Keywords: lipoedema; obesity
MeSH Terms: conditions — Lipedema; Obesity | interventions — Muscle Strength; Body Mass Index

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- patient with lipoedema (Active Comparator): Lipedema group:
  * diagnosed with lipedema following the criteria of Wold
  * women
  * age ≥ 18 years
  clinimetrics: volume, muscle strength, physical condition, BMI
  Interventions: Other: volume, muscle strength, physical condition, BMI
- patients with obesity (Active Comparator): Obesity group:
  * BMI ≥ 30
  * women
  * age ≥ 18 years
  clinimetrics: volume, muscle strength, physical condition, BMI
  Interventions: Other: volume, muscle strength, physical condition, BMI

INTERVENTIONS:
Other: volume, muscle strength, physical condition, BMI — phys. condition, muscle strength, volumetry, BMI

SUMMARY:
The diagnosis of lipoedema and obesity are often mixed up, unclear stated and often there is a misdiagnosis. The primary aim is to investigate whether there is a difference in muscle strength between women with lipedema and women with obesity. The secondary aim is to investigate whether there is a difference in physical fitness between women with lipedema and women with obesity.

DETAILED DESCRIPTION:
Lipedema is a genetically mediated disorder of adipose tissue that occurs exclusively in women. Lipedema is an under-recognized condition, often misdiagnosed as lymfedema or dismissed as simple obesity. The diagnosis of lipedema is a clinical diagnosis and may be challenging to determine among patients who are obese. Measurements of muscle strength and physical fitness may give more clarity to differentiate between lipedema and obesity. This may lead to improvements in the criteria of diagnosing lipedema. The research question of the study is: Is there a difference in muscle strength between adult women with lipedema and adult women with obesity?

In this study 40 patients will be studied; 20 patients in every group. Besides the general data as length, weight, age, abdominal circumference, volume of the legs additional muscle strength and physical fitness of women with lipedema and women with obesity will be measured and analysis.

This study doesn't involve a negligible risk for participants. The study will not have direct benefit for the participants, but may be useful in giving more clarity in defining the phenotype for patients with lipedema.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

Lipedema group:

* diagnosed with lipedema following the criteria of Wold et al3
* women
* age ≥ 18 years

Obesity group:

* BMI ≥ 30
* women
* age ≥ 18 years

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

Lipedema group:

- none

Obesity group:

- an obesity intervention with physical training in the ≤12 months prior to the measurement

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-12; Primary Completion 2013-06 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
The main determinant of this study is a muscle strength test of the Quadriceps muscle of the left and right leg measured with the MircoFET. | June 2013
  Muscle strength will be measured with the MicroFET. This test is performed when de patient is sitting. The patient is instructed to perform knee extension three times for each leg. The test result is de average score of each leg. The MicroFET has been shown to be a valid measurement with the break-method.14,15 Schaubert et al.15 and Bohannon et al.14 looked at the reliability of MicroFET measurements and found a good Intraclass Correlation Coefficient (ICC) values of 0.807-0.97115 and ICC>.097014 respectively. The test procedure of the break-method is described in Appendix 1).

SECONDARY OUTCOMES:
walking capacity | June 2013
  After performing the muscle strength test, the participants will be asked to perform a test for physical fitness, knowing the Six Minute Walk Test (6MWT). Walking capacity will be measured with the 6MWT. This standardized test is performed on a 30 meters course where every five meter is marked. The patient will be instructed to cross a maximum distance in six minutes with a possibility to stop or rest if necessary.16 The result is the walking distance in meters (m) after six minutes (with five meter exactness). The 6MWT is a good test for functional activity. De walking distance performed with the 6MWT gives a good sight in the amount of activities in daily living (ADL) of the performer.17 Rjeski et al.17 found a good validity and correlation with the VO2max (r=0.64) for participants with chronic obstructive pulmonary disease (COPD). The test-retest reliability of this test is good (ICC 0.94).18

CONTACTS AND LOCATIONS:
Overall Officials: RJ Damstra, MD PhD, Principal Investigator — Nij Smellinghe Hospital
Locations (1):
- Expert Center for Lymphovascular Medicine Nij Smellinghe Hospital, Drachten, Provincie Friesland, Netherlands

REFERENCES:
- See also: General website form the Nij Smellinghe hospital — http://www.nijsmellinghe.nl
- See also: The foundation related to the expert centre organizing research — http://www.slcn.nl